CLINICAL TRIAL: NCT02064153
Title: Potential of Manipulating the Dialysate Temperature for Prevention of Intra-dialytic Hypotensive Episodes in Maintenance Hemodialysis Patients
Brief Title: Studying the Effect of Dialysate Temperature on Toxin Removal and Hypotension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National University Hospital, Singapore (Other)
Collaborators: National University of Singapore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: DSRB 2013/1950
Record Dates: First submitted 2014-02-13; First posted 2014-02-17 (Estimated); Last update posted 2015-04-03 (Estimated); Status verified 2015-04

CONDITIONS: Dialysis Amyloidosis; Hypotension
Keywords: Dialysate temperature; Spent dialysate; Toxin removal; Intra-dialytic hypotension; Inter-compartmental resistance
MeSH Terms: conditions — Hypotension

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cool dialysate (Active Comparator): Recruited study subject undergoes cool dialysate (35.5ºC) session.
  Interventions: Procedure: Cool dialysate
- Warm dialysate (Active Comparator): Recruited study subject undergoes warm dialysate (37ºC) session.
  Interventions: Procedure: Warm dialysate

INTERVENTIONS:
Procedure: Cool dialysate — Each recruited patient undergoes a cool dialysate session ( 35.5ºC) and a warm dialysate session (37ºC). The sessions are minimum a week apart to remove the carryover effect.
  Other Names: Cool dialysate at 35.5ºC; Warm dialysate at 37ºC
  Arms: Cool dialysate
Procedure: Warm dialysate — All recruited patients will undergo two study sessions - Cool dialysis (35.5ºC) and Warm dialysis (37ºC)
  Other Names: Warm dialysate at 37ºC
  Arms: Warm dialysate

SUMMARY:
Hemodialysis (HD) is widely used treatment for end stage renal diseases (ESRD) patients. The chief aims of HD are solute and fluid removal. Decades of practice have improved HD care, but more can be done to improve morbidity and mortality. Enhancing toxin removal is an important consideration for improved patient outcomes. Also, decreasing the incidence of intra-dialytic hypotensive (IDH) episodes (dominant in Singapore patient cohort) can significantly reduce associated morbidities and mortality. A simple maneuver for clinicians is the dialysate temperature. Literature suggests that a lower dialysate temperature (35ºC) results in reduced hypotensive episodes by vasoconstriction. Conversely, higher dialysate temperature resulting in higher blood temperature decreases the peripheral resistance, leading to increased toxin removal, but may cause IDH episodes partly due to vasodilation. Optimal manipulation of the dialysate temperature is therefore primary handles to obtain the improved patient outcomes. In this study, the effect of dialysate temperature (cool vs. warm dialysate) on toxin removal will be studied. In both the interventions, outcome measure will be patient hemodynamic response and amount of toxins removed. The spent dialysate will be collected to study the quantum of toxin removed.

DETAILED DESCRIPTION:
Cool dialysate, by vasoconstriction, is simple maneuver to control and/or prevent incidence of intra-dialytic hypotension (IDH). During dialysis fluid is continuously removed. IDH occurs when plasma refilling rate is smaller than the set ultra-filtration rate. When plasma refiling rate is small, continuous fluid removal bring patient to the threshold state where patient does not have sufficient fluid in central compartment. This leads to the cascade of events, viz., low blood pressure, muscle cramps, dizziness, being first few manifestation. To minimize the occurrence of such events, clinicians often prescribe cool dialysate resulting in vasoconstriction, which ensures sufficient fluid volume in central body compartment so that continuous fluid loss does not impact patient hemodynamics severely.

It is important to note that vasoconstriction may also inhibit the toxin movement from remote peripheral compartments to central blood compartment, and thus less toxin will be removed. On the other hand warm dialysate leading to vasodilation will mobilize the toxins in remote peripheral compartments and increase the toxin influx in central blood compartment. Few researchers have investigate the effect of dialysate temperature on urea removal, but urea is not a true marker of toxin milieu. In this pilot clinical research, we will compare the effect of dialysate temperature on removal of both small and large sized uremic toxins. Our objective is not to study the effect of dialysate temperature on incidence of IDH, so we will recruit subjects who are stable on dialysis and have no prior history of IDH episodes.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients male or female (Age > 21 years, < 70 years)
2. Minimum dialysis vintage of 3 months
3. Stable on hemodialysis
4. Blood access capable of delivering the blood flow rate greater than 250 mL/min

Exclusion Criteria:

1. History of recurring or persistent hypotension in past 1 month
2. Pregnant woman
3. Severely hypertensive patients (Systolic blood pressure > 180 mmHg and/or Diastolic blood pressure > 115 mmHg)
4. Severely hypotensive patients (Systolic blood pressure < 100 mm Hg and/or Diastolic blood pressure < 60 mmHg)
5. Paradoxically hypertensive patients whose BP increases by more than 20% of baseline during dialysis (during past 1 month)
6. History of recent myocardial infarction or unstable angina (within past 6 months)
7. Significant valvular disease, i.e. severe aortic stenosis and moderate-severe mitral regurgitation
8. Patients with end stage organ disease e.g. chronic obstructive pulmonary disease (COPD), recent or debilitating cerebrovascular attack (CVA)
9. Patient with recent stroke (within past 6 months)
10. History of known arrhythmia
11. Participation in another clinical intervention trial
12. Unable to consent

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2013-07; Primary Completion 2014-03 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Quantify toxin removal based on spent dialysate | 1 month
  Collect the whole dialysate and measure the toxin concentration. This will provide the amount of toxin removed during study session. Compare the removed toxin mass for cool vs warm dialysate session.

SECONDARY OUTCOMES:
Monitoring of physiological changes | 1 month
  Cool dialysate may lead to stability of patient, but may also result in chilling sensation during dialysis. On the other hand, warm dialysate may cause intra-dialytic hypotensive episode. In both sessions, patient physiological changes will be monitored.

CONTACTS AND LOCATIONS:
Overall Officials: Titus Lau, MD, Study Director — National University Hospital, Singapore; Vaibhav Maheshwari, PhD, Principal Investigator — National University of Singapore
Locations (1):
- SLF Dialysis Center, National University Hospital, Singapore, SGN, Singapore

REFERENCES:
- [Background] Kaufman AM, Morris AT, Lavarias VA, Wang Y, Leung JF, Glabman MB, Yusuf SA, Levoci AL, Polaschegg HD, Levin NW. Effects of controlled blood cooling on hemodynamic stability and urea kinetics during high-efficiency hemodialysis. J Am Soc Nephrol. 1998 May;9(5):877-83. doi: 10.1681/ASN.V95877. PMID 9596086
- [Derived] Maheshwari V, Lau T, Samavedham L, Rangaiah GP. Effect of cool vs. warm dialysate on toxin removal: rationale and study design. BMC Nephrol. 2015 Feb 27;16:25. doi: 10.1186/s12882-015-0017-5. PMID 25885180
- See also: Effects of controlled blood cooling on hemodynamic stability and urea kinetics during high-efficiency hemodialysis — http://www.ncbi.nlm.nih.gov/pubmed/9596086
- See also: A regional blood flow model for β2-microglobulin kinetics and for simulating intra-dialytic exercise effect — http://www.ncbi.nlm.nih.gov/pubmed/21877220